CLINICAL TRIAL: NCT06386120
Title: Respiratory Function Monitoring of Patients With Chest Blunt Injury With Mechanical Ventilation
Brief Title: Respiratory Function Monitoring of Mechanical Ventilation in Patients With Chest Blunt Injury
Status: Not yet recruiting | Type: Observational
Sponsor: Peking University People's Hospital (Other)
Responsible Party: Principal Investigator, Li Shu, associate professor, Peking University People's Hospital
Other Study IDs: 2024-z033
Record Dates: First submitted 2024-04-24; First posted 2024-04-26 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Lung Contusion
Keywords: chest contusion; lung contusion; electrical impedance tomography; pulmonary perfusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- EIT-PEEP group: The PEEP titration guided by EIT, decided by the responsible attending physician
  Interventions: Other: PEEP setting strategy
- Table-PEEP group: The PEEP setting with low FiO2-PEEP table, decided by the responsible attending physician
  Interventions: Other: PEEP setting strategy

INTERVENTIONS:
Other: PEEP setting strategy — The attending physician selects different PEEP setting strategies

SUMMARY:
The goal of this observational study is to learn about EIT in observing the application of lung protective ventilation strategies in patients with pulmonary contusion, particularly the impact on pulmonary ventilation blood flow ratio, oxygen, and condition. The main question it aims to answer is:

Can lung protective ventilation strategies improve respiratory function in patients with severe chest contusion? We will collect clinical data of participants who already taking lung protective ventilation strategies as part of their regular medical care.

DETAILED DESCRIPTION:
Trauma is the leading cause of death among middle-aged and young people in China, with over 25% of patients dying from chest trauma. The incidence of pulmonary contusion in severe chest trauma is over 70%, and it is an important cause of respiratory failure and even death in patients. The occurrence of pulmonary contusion and respiratory failure in patients with chest contusion is a dynamic process, and Regional inhomogeneities of the damaged lung should be taken into consideration to develop improved ventilation strategies. Currently, there is no ideal monitoring method to evaluate the severity of injury, and guide the ventilation strategies. Electrical impedance tomography (EIT) is a non-invasive, radiation-free imaging technique. It measures regional lung ventilation and aeration distribution by means of changes in electrical potentials at the skin surface of the chest wall during breathing cycles, which has been proven to have good practicality in patients with non-invasive ARDS and pulmonary embolism. In this study, we aim to characterize the physiologic effects of positive end expiratory pressure (PEEP) on key mechanisms of regional lung protection, namely: recruitment, reduced atelectrauma, and improved ventilation-perfusion matching, by CT scan and EIT

ELIGIBILITY:
Inclusion Criteria:

* Patients with severe chest contusion admitted to the intensive care unit (ICU);
* Abbreviated Injury Scale (AIS) ≥ 3 and/or Blunt Pulmonary Contusion 18 score (BPC18) ≥ 3;
* Age range from 18 to 90 years old;
* Mechanical ventilation;
* Stay in the ICU for less than 12 hours.

Exclusion Criteria:

* Perinatal women;
* Expected to be mechanically ventilated for less than 48 h;
* Expected duration of stay in the ICU is less than 24 hours;
* There are contraindications for the use of EIT (pacemaker implantation, local skin wounds after chest surgery, etc.);
* Accept extracorporeal membrane oxygenator;
* Mechanical ventilation>7 days;
* Confirmed ventilator-associated pneumonia;
* Pneumothorax without drainage or presence of subcutaneous emphysema.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The cohort will be selected from a tertiary hospital
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2026-05 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
ventilation blood flow ratio | through study completion, an average of 1 year
  ventilation blood flow ratio of lung

SECONDARY OUTCOMES:
oxygenation index | through study completion, an average of 1 year
  oxygenation index of participant
28-day mortality | through study completion, an average of 1 year
  28-day mortality
Mechanical ventilation-free from day 1 to 28 | through study completion, an average of 1 year
  Mechanical ventilation-free from day 1 to 28
Length of ICU stay | through study completion, an average of 1 year
  Length of ICU stay
Length of hospital stay | through study completion, an average of 1 year
  Length of hospital stay
The rate of successful weaning | through study completion, an average of 1 year
  the absence of the requirement for ventilatory support, without reintubation, a cardiac arrest event, or mortality within 48h after extubating or withdrawal

CONTACTS AND LOCATIONS:
Overall Officials: Shu Li, doctor, Principal Investigator — Peking University People's Hospital

IPD SHARING:
Plan to Share IPD: Yes
all collected IPD, all IPD that underlie results in a publication
Supporting Information: Study Protocol, SAP, ICF
Time Frame: starting 1 year after publication
Access Criteria: The data used and/or analyzed during the current study are available from the Investigator on reasonable request.